CLINICAL TRIAL: NCT03703817
Title: TREATMENT SATISFACTION COMPARISON IN RHEUMATOID ARTHRITIS PATIENTS BETWEEN TOFACITINIB CITRATE AND ADALIMUMAB, EACH USED IN RHEUMATOID ARTHRITIS TREATMENT
Brief Title: Rheumatoid Arthritis Satisfaction Outcome Research
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: A3921304; RA SATISFACTION (Other: Alias Study Number)
Record Dates: First submitted 2018-06-22; First posted 2018-10-12 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- tofacitinib citrate users: patients who have been using tofacitinib citrate for 6 months or more and less than 2 year in RA patients
- adalimumab users: patients who have been using adalimumab for 6 months or more and less than 2 year in RA patients

SUMMARY:
RA satisfaction OR: This study aim to compare treatment satisfaction and quality of life between patients who have been using tofacitinib citrate and patients who have been using adalimumab for 6 months or more and less than 2 year in RA treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
RA satisfaction OR: This study aim to compare treatment satisfaction and quality of life between patients who have been using tofacitinib citrate and patients who have been using adalimumab for 6 months or more and less than 2 year in RA treatment of rheumatoid arthritis.

Study design: Non-interventional, multi-centers, cross-sectional study

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years or older
2. Patients diagnosed with RA
3. Treatment groups:

1) Tofacitinib citrate users: Patients currently on treatment with tofacitinib citrate in RA therapy for 6 months or more 2) Adalimumab users: Patients currently on treatment with adalimumab in the RA therapy for 6 months or more 4. Reading and writing with enough proficiency to complete assessment instruments in Korean

Exclusion Criteria:

1. Patients currently on tofacitinib citrate or adalimumab for 2 year or more
2. Patients taking Azathioprine and cyclosporine
3. Patients participating in other drug interventional study
4. Patients who have been treated with bDMARDs except Rheumatoid arthritis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is RA patients who have been using tofacitinib citrate or adalimumab for 6 months or more and less than 2 year in RA treatment at participating institution
Sampling Method: Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- South Korea (23):
  - Kyung Hee University Hospital at Gangdong / Rheumatology, Seoul, Gangdong-gu
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Wonkwang University Hospital / Division of Rheumatology, Iksan, Jeonlabuk-do
  - Ajou University Hospital, Department of Rheumatology, Suwon, Kyeongki-do
  - Eulji University Hospital, Daejeon, Republic of Korea
  - Asan Medical Center, Songpa-gu, Seoul
  - Hallym University Sacred Heart Hospital/Rheumatology, Internal Medicine, Anyang
  - Inje University Busan Paik Hospital, Department of Internal Medicine, Busan
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Daegu Catholic University Medical Center, Department of Rheumatology, Daegu
  - Gacheon Medical School Gil Medical Center, Rheumatology, Internal Medicine, Incheon
  - Pusan National University Hospital, Pusan
  - Dong-A University Hospital, Pusan
  - Hanyang University Seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Hanyang University Hospital, Department of Rheumatology, Seoul
  - Catholic University of Korea, Kangnam St. Mary's Hospital, Seoul
  - Konkuk University Hospital, Department of Rheumatology, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Kim SK, Lee SH, Sun J, Lee SH, Jeon JY, Yoo HJ, Choe JY. Comparisons of treatment satisfaction and health-related quality of life in patients with rheumatoid arthritis treated with tofacitinib and adalimumab. Arthritis Res Ther. 2023 Apr 27;25(1):68. doi: 10.1186/s13075-023-03047-1. PMID 37106411
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921304

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study data was collected from participants who had been using tofacitinib citrate or adalimumab for 6 months or more and less than 2 years for rheumatoid arthritis (RA) treatment. Data was collected and analyzed from 2-July-2018 to 12-March-2020 (approximately 20 months), for comparing treatment satisfaction and quality of life between the 2 treatment groups.
Groups:
- Tofacitinib Citrate: Participants who had been using tofacitinib citrate for more than 6 months or more and less than 2 years for RA treatment were included in the group.
- Adalimumab: Participants who had been using adalimumab for more than 6 months or more and less than 2 years for RA treatment were included in the group.
Period: Overall Study
Arm/Group | Tofacitinib Citrate | Adalimumab
Started | 288 | 133
Completed | 281 | 129
Not Completed | 7 | 4
Not completed — Not meeting eligibility criteria | 7 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who satisfied the inclusion criteria and were registered for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Citrate | Adalimumab | Total
Number analyzed (Participants) | 281 | 129 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.473 (12.098) | 51.450 (12.176) | 53.522 (12.189)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 115 | 356
  Male | 40 | 14 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Version 1.4
Description: TSQM version 1.4: participant rated 14 items with 4 domains. Scores for item 1 to 3, 9 to 11 and 14 ranged from 1=extremely dissatisfied to 7=extremely satisfied. Items 5 to 8, 12, 13 ranged from 1=extremely dissatisfied to 5=not at all dissatisfied. Item 4 was scored as: 0=No, 1=Yes. Effectiveness measured as ([{sum of item 1 to 3} - 3]/18)*100; if 1 question (Q) was missing: ([{sum of item 1 to 3} -2]/12)*100. Side-effect measured as if item 4=No, score=100; if not then ([{sum of item 5 to 8} -4]/16)*100; if 1 Q was missing: ([{sum of item 5 to 8} -3]/12)*100. Convenience measured as ([{sum of item 9 to 11} -3]/18)*100; if 1 Q was missing: ([{sum of item 9 to 11} - 2]/12)*100. Global satisfaction as ([{sum of item 12 to 14} -3]/14)*100; if item 12 or 13 was missing: ([{sum of item 12 to 14} -2]/10)*100; if item 14 was missing: ([{sum of item 12 and 13} -2]/8)*100. All domains had scale of 0 (no satisfaction) to 100 (best level of satisfaction), higher score=greater satisfaction.
Time Frame: Day 1 (during approximately 20 months of data collection and observation)
Population: The propensity score method (greedy matching method) was used in analysis of the outcome measure. The purpose of the propensity score was to create conditions similar to those of randomized trials by balancing the covariates in participants between the groups. It reduces multidimensional covariates into a one-dimensional score. Here, 'Overall Number of Participants Analyzed' signifies number of participant evaluable for this outcome measure derived from propensity score method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Citrate | Adalimumab
Number analyzed (Participants) | 139 | 92
units on a scale
  Effectiveness | 62.271 (13.301) | 64.191 (13.315)
  Side effects | 93.390 (16.668) | 96.603 (11.625)
  Convenience | 68.785 (13.349) | 64.946 (12.845)
  Global satisfaction | 56.680 (15.412) | 59.860 (15.558)
Statistical Analysis 1: Comparison: Tofacitinib Citrate vs Adalimumab; Test type: Superiority — Effectiveness: Multivariate analysis was used to control and remove the possible influence of the independent variables (demographic and clinical characteristics); p = 0.3648, Linear mixed model
Statistical Analysis 2: Comparison: Tofacitinib Citrate vs Adalimumab; Test type: Superiority — Side effect: Multivariate analysis was used to control and remove the possible influence of the independent variables (demographic and clinical characteristics); p = 0.1395, Conditional logistic regression
Statistical Analysis 3: Comparison: Tofacitinib Citrate vs Adalimumab; Test type: Superiority — Convenience: Multivariate analysis was used to control and remove the possible influence of the independent variables (demographic and clinical characteristics); p = 0.0349, Linear mixed model
Statistical Analysis 4: Comparison: Tofacitinib Citrate vs Adalimumab; Test type: Superiority — Global satisfaction: Multivariate analysis was used to control and remove the possible influence of the independent variables (demographic and clinical characteristics); p = 0.1546, Linear mixed model

2. Secondary Outcome: European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Index Score
Description: EQ-5D-3L assess health-related quality of life. It has 5 dimensions: mobility (M), self-care (SC), usual activities (UA), pain/discomfort (PD) and anxiety/depression (AD). Each dimension has 3 levels. For mobility, self-care and usual activities: 1= no effects, 2= sometimes affected, 3= very affected. For pain/discomfort and anxiety/depression: 1= none, 2= sometimes, 3= often. EQ-5D-3L index was calculated using formula = 1 - (0.0081 + [0.1140 * M2 + 0.6274 * M3 + 0.0572 * SC2 + 0.2073 * SC3 + 0.0615 * UA2 + 0.2812 * UA3 + 0.0581 * PD2+ 0.2353 * PD3 + 0.0675 * AD2 + 0.2351 * AD3]). In this formula, abbreviated form for dimension is followed by level, for example M2 = mobility level 2. Values were set to 1 if level was 2 or 3 for M2, SC2, UA2, PD2, AD2 or M3, SC3, UA3, PD3, AD3 respectively, else set to 0. Total score ranged from -0.27 to 1. Higher scores indicate better health.
Time Frame: Day 1 (during approximately 20 months of data collection and observation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Citrate | Adalimumab
Number analyzed (Participants) | 139 | 92
units on a scale | 0.812 (0.146) | 0.808 (0.134)
Statistical Analysis 1: Comparison: Tofacitinib Citrate vs Adalimumab; Test type: Superiority — Multivariate analysis was used to control and remove the possible influence of the independent variables (demographic and clinical characteristics); p = 0.1602, Conditional logistic regression model

3. Secondary Outcome: European Quality of Life-Visual Analogue Scale (EQ-VAS) Score
Description: EQ-VAS is a standardized tool for measuring overall health. EQ-VAS recorded the participant's self-rated health on a vertical, VAS on a scale ranging from and 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicated better health state.
Time Frame: Day 1 (during approximately 20 months of data collection and observation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Citrate | Adalimumab
Number analyzed (Participants) | 139 | 92
units on a scale | 65.403 (19.974) | 65.668 (19.554)
Statistical Analysis 1: Comparison: Tofacitinib Citrate vs Adalimumab; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9921, Linear mixed model

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last administration of tofacitinib citrate or adalimumab (during approximately 20 months of data collection and observation)
Description: Full analysis set included all participants who satisfied the inclusion criteria and were registered for the study.
Arm/Group | Tofacitinib Citrate | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/281 | 0/129
Other Adverse Events (participants affected / at risk) | 2/281 | 0/129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Citrate (N=281) | Adalimumab (N=129)
Viral infection (Infections and infestations) | 1 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03703817/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03703817/SAP_001.pdf